CLINICAL TRIAL: NCT02198443
Title: Prophylaxis for HIV-1: Tenofovir/Emtricitabine (Truvada ®) + Lopinavir/Ritonavir (Kaletra ®) vs Tenofovir/Emtricitabine/Cobicistat/Elvitegravir (Stribild ®). Prospective, Randomized, Open.
Brief Title: Comparison of Two Combinations in Antiretroviral Post-Exposure Prophylaxis for HIV-1: Tenofovir/Emtricitabine (Truvada ®) + Lopinavir/Ritonavir (Kaletra ®) vs Tenofovir/Emtricitabine/Cobicistat/Elvitegravir (Stribild ®). Prospective, Randomized, Open.
Acronym: STRIB-PEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, project manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STRIB-PEP
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2014-07

CONDITIONS: HIV
MeSH Terms: interventions — Tenofovir; Emtricitabine; Ritonavir; lopinavir-ritonavir drug combination; elvitegravir; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenofovir+emtricitabine (Active Comparator)
  Interventions: Drug: Tenofovir + emtricitabine (Truvada),+lopinavir/ritonavir (Kaletra)
- Elvitegravir/cobicistat/emtricitabine/Tenofovir-Disoproxil (Experimental)
  Interventions: Drug: elvitegravir/cobicistat/emtricitabine/Tenofovir-Disoproxil

INTERVENTIONS:
Drug: Tenofovir + emtricitabine (Truvada),+lopinavir/ritonavir (Kaletra) — (TRUVADA) film-coated 200/245 mg tablet / day tablets (Kaletra) film-coated 200/50 mg tablets twice / day tablets
  Arms: Tenofovir+emtricitabine
Drug: elvitegravir/cobicistat/emtricitabine/Tenofovir-Disoproxil — Film-coated tablets of 150 mg of elvitegravir, cobicistat 150 mg, 200 mg of emtricitabine and 245 mg of tenofovir disoproxil. One tablet once / day.
  Other Names: (Stribild)
  Arms: Elvitegravir/cobicistat/emtricitabine/Tenofovir-Disoproxil

SUMMARY:
The main objective of this study is to compare the tolerability and adherence to a new drug regimen of post-exposure prophylaxis (PEP) for HIV,

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Have been exposed to HIV, non-occupational and meets the requirements of current recommendations to start with three antiretroviral drugs PEP
* that adequately informed consent in writing to participate in the study and undergo testing and exploration that entails

Exclusion Criteria:

* pregnant women, lactating, or those intend become pregnant during the study period.
* subjects who are known or suspected case presents the source resistors to one of the drugs of the pattern of study
* contraindicated treatment with the study drugs, or products under investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-06-06 (Actual); Primary Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who leave the initial treatment of post-exposure prophylaxis (PEP) for HIV for any reason | Twenty Eigth days
  A subject is considered to abandon treatment if within 28 days
  * dies
  * Do not come to visit week 4
  * changed or discontinued study treatment.

SECONDARY OUTCOMES:
Incidence of clinical adverse events and / or laboratory alterations. | twenty-four weeks
Proportion of patients who discontinued treatment due to toxicity or intolerance in each of the treatment arms at 24 weeks follow-up | twenty four weeks
degree of adhesion during the treatment period | twenty eight days
  Measured by pill count and patient adherence questionnaire
time to loss of adherence to TARV | twenty eight days
Proportion of patients with seroconversion in both treatment arms at 24 weeks follow-up. | twenty four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Felipe García, MD, Principal Investigator — Hospital clínic y provincial de Barcelona
Locations (1):
- Hospital clínico y provincial de Barcelona, Barcelona, Barcelona, Spain